CLINICAL TRIAL: NCT01149252
Title: Determination of the Efficacy and Safety of Psoralait Versus Placebo in the Treatment of Psoriasis.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties arouse in recruiting new patients
Sponsor: Trima, Israel Pharmaceutical Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Psoriasis
Record Dates: First submitted 2010-06-20; First posted 2010-06-23 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psoralait (Placebo Comparator)
  Interventions: Other: Psoralait; Other: Placebo cream.

INTERVENTIONS:
Other: Psoralait — Cream to be used as instructed.
Other: Placebo cream. — Cream to be used as instructed

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a new product, Psoralait, as compared to a placebo in the treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been clinically diagnosed as suffering from psoriasis and are or aren't scheduled for Narrow Band Ultraviolet B (UVB)phototherapy of affected areas,excluding face and genitalia.

Exclusion Criteria:

* Women who are pregnant, lactating, planning to become pregnant, or women of child-bearing potential who have not successfully been using the same medically acceptable contraceptive methods over the previous 3 months, e.g., oral contraceptive agents, intrauterine device (IUD) and barrier method plus spermicide.
* Use of topical anti psoriatic therapy (including topical retinoids, corticosteroids, or vitamin D analogs) on the areas to be treated within 2 weeks prior to the beginning of the study.
* Received systemic biologic therapy to treat psoriasis (for example: alefacept, etanercept, infliximab, adalimumab) within 12 weeks prior to the beginning of the study.
* Received systemic psoriasis therapy (for example: methotrexate, cyclosporine, systemic corticosteroids, retinoids such as acitretin) within 4 weeks prior to the beginning of the study.
* Received phototherapy (including laser), photo chemotherapy or climatotherapy within 4 weeks prior to the beginning of the study.
* Recent history (within past 12 months) of alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1.5 oz distilled spirits).
* History of noncompliance to medical regimens or unwilling to comply with the study protocol.
* Participation in an investigational drug study within 30 days prior to the beginning of the study.
* Serious or unstable medical or psychological conditions that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI). | After four weeks of treatment.

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI). | After four weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Phototherapy and Dermatology Day Care Center, Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel